CLINICAL TRIAL: NCT06102889
Title: GUIDING MULTI-MODAL THERAPIES AGAINST MINIMAL RESIDUAL DISEASE BY LIQUID BIOPSIES
Acronym: GUIDEMRD
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Aarhus University Hospital (Other); Centre Hospitalier Universitaire de Nice (Other); Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other); Medical University of Graz (Other); Centre Hospitalier Régional Universitaire Montpellier (Other)
Responsible Party: Principal Investigator, Matthias Löhr, Professor of Gastroenterology & Hepatology, Karolinska University Hospital
Other Study IDs: GUIDE.MRD-02-PDAC
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Liquid biopsy
MeSH Terms: interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for circulating tumour DNA (ctDNA), exosomes, proteomics, metabolomics, and circulating tumour cells (CTC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: liquid biopsy — Taking blood samples (liquid biopsy) for multiple analysis in genomics, proteomics, and metabolomics

SUMMARY:
The overall objective of this study is to confirm that ctDNA detected after curative intended treatment for PDAC is a marker of residual disease and for risk-of-recurrence, and applicable in clinical practice.

Primary objective To confirm that ctDNA analyses performed after PDAC treatment can identify patients with a high risk-of-recurrence.

Specifically, we want to determine the association between disease-free survival (DFS) and ctDNA detection status after (1) curative-intended surgery and (2) adjuvant chemotherapy.

DETAILED DESCRIPTION:
The study will prospectively enroll patients who undergo potentially curative surgery for PDAC. The intervention is repeated blood sampling at pre-defined time points.

Patient identification Patients with PDAC are screened for eligibility by the involved physicians based on the protocol of the multidisciplinary tumor board (MDT). The screening will be done based on the electronic health record in the electronic journal (at present, for example, Take Care). The National Health Record may be accessed for some patients to complete the record.

Patient recruitment and informed consent The involved physicians screen patients meeting the inclusion criteria specified below. Eligible patients are approached in person or initially by phone, after they have been informed about the diagnosis and the planned surgery. Patients are given written and oral information about the project by a trained research nurse or by an involved physician. Informed consent will be obtained before the beginning of any study-related procedures.

The signed and dated consent forms are scanned into the project's electronic database and stored physically in a locked space.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic ductal adenocarcinoma, according to the assessment of the MDT.
* Age 18 years or older.
* Patient able to understand and sign written informed consent in Swedish.
* Scheduled for curative intent surgical resection.

Exclusion Criteria:

* Hereditary pancreatic cancer.
* Verified distant metastases.
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits and/or otherwise considered by the Investigator to be unlikely to complete the study.
* Other cancers (excluding prior pancreatic cancer or skin cancer other than melanoma) within 3 years from eligibility screening.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with histologically verified pancreatic adenocarcinoma (from surgically removed tumour tissue = ground truth) regardless of their ability to receive SOC adjuvant chemotherapy or not (observation only - due to pre-existing medical conditions), regardless of type of chemotherapy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pancreatic cancer | 1 month - 24 months after surgical resection of the tumor
  Occurence of a "positive" biomarker or markers after adjuvant chemotherapy prior to clinically overt recurrence.

SECONDARY OUTCOMES:
Effect of standard-of-care (SOC) chemotherapy on biomarker(s) | 1 month - 24 months after surgical resection of the tumor
  Disappearance or re-occurence of a "positive" biomarker or markers after adjuvant chemotherapy prior to clinically overt recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Lindbjerg Andersen, MD, Study Director — Aarhus University Hospitsl
Locations (1):
- Gastrocentrum, KarolinskaUniversity Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
After completion of the study, the SAB and study group to decide whether to share the results on a group level, i.e. anonymously